CLINICAL TRIAL: NCT02767414
Title: A Prospective Multi-centre Study of the Ellume® Respirio Flu Test and the Ellume® eLab Flu Test Performance Versus Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) for the Rapid Detection of Influenza A/B
Brief Title: Validation of the Ellume® Respirio Flu Test and the Ellume® eLab Flu Test for the Rapid Identification of Influenza A/B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellume Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RESP16001
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Influenza A; Influenza B
MeSH Terms: interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respirio Flu Test and eLab Flu Test (Experimental): Upper respiratory tract samples from participants will be tested with:
  Respirio Flu Test; eLab Flu Test; and Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)
  Interventions: Device: Respirio Flu Test; Device: eLab Flu Test; Device: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)

INTERVENTIONS:
Device: Respirio Flu Test — The Respirio Flu Test is a rapid in vitro diagnostic test for the detection of influenza A or influenza B in nasal secretions. The Respirio Flu Test is designed to be simple to use and generates a result within 20 minutes.
Device: eLab Flu Test — The eLab Flu Test is an in vitro diagnostic test intended to be used at point-of-care for the detection of influenza A or influenza B in nasopharyngeal swab samples. The eLab Flu Test generates a result within 10 minutes.
Device: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) — Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) is a molecular diagnostic technique for the detection and identification of influenza viruses, both for clinical samples and isolates. The reverse transcriptase polymerase chain reaction (RT-PCR) allows template viral RNA to be reverse transcribed producing complementary DNA (cDNA) which can then be amplified and detected.

SUMMARY:
The primary purpose of this study is to validate the sensitivity and specificity of the Respirio Flu Test and the eLab Flu Test in detecting Influenza A as compared to the gold standard for detection, Reverse Transcriptase Polymerase Chain Reaction (RT-PCR).

The secondary aims are to:

Validate the sensitivity and specificity of the Respirio Flu Test and the eLab Flu Test in detecting Influenza B as compared to the gold standard for detection, Reverse Transcriptase Polymerase Chain Reaction (RT-PCR); Evaluate the correct interpretation of the Respirio Flu Test by subjects with influenza-like symptoms; Evaluate the subjects' satisfaction with the convenience, comfort and ease of use of the Respirio Flu Test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 1 year;
* Rhinorrhea;
* ≤ 5 days from onset of influenza-like illness symptoms;
* Subject (or parent/legal guardian) capable and willing to give informed consent/assent;
* Subject (or parent/legal guardian) able to read and write English.

Exclusion Criteria:

* Has undergone treatment with antivirals within the previous 7 days;
* Has been vaccinated by means of an influenza nasal spray/mist vaccine within the previous 7 days;
* Recent craniofacial injury or surgery, including surgery to correct deviation of the nasal septum, within the previous 6 months;
* Currently enrolled in another clinical trial or used any investigational device within 90 days preceding informed consent;
* Has had prior exposure to the Respirio Flu Test or eLab Flu Test.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Of participants positive for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza A by Respirio Flu Test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza A by eLab Flu Test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza A by Respirio Flu Test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza A by eLab Flu Test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.

SECONDARY OUTCOMES:
Of participants positive for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza B by Respirio Flu Test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza B by eLab Flu Test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza B by Respirio Flu Test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants negative for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza B by eLab Flu Test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Percent of participants who correctly interpret result of Respirio Flu Test. | Day 1
  Agreement between trained staff and participants. Report as a percentage of participants with 95% confidence limits.
Scores from questionnaire to assess ease of use, comfort and convenience of Respirio Flu Test. | Day 1
  The ease of use questionnaire will provide total number of responses to each question and the percentage of participants selecting each response (on a 5 point Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Noel Cranswick, Principal Investigator — Australian Paediatric Pharmacology Research Unit, Royal Children's Hospital; James Pollard, Principal Investigator — Barwon Health - Geelong; Paul Griffin, Principal Investigator — Mater Hospital - Brisbane; Stephen Windley, Principal Investigator — Doctors@Carindale; Luke Katahanas, Principal Investigator — Capalaba Medical Centre; Bernardine McKellar, Principal Investigator — Red Hill Doctors Surgery; Evan Jones, Principal Investigator — University of Sunshine Coast Clinical Trials Centre
Locations (7):
- Australia (7):
  - Red Hill Doctors Surgery, Brisbane, Queensland
  - Mater Hospital - Brisbane, Brisbane, Queensland
  - Doctors@Carindale, Brisbane, Queensland
  - Capalaba Medical Centre, Redland, Queensland
  - Clinical Trials Centre - University of the Sunshine Coast, Sippy Downs, Queensland
  - Barwon Health - Geelong, Geelong, Victoria
  - The Royal Children's Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No